CLINICAL TRIAL: NCT03918629
Title: A PHASE 3, RANDOMIZED OBSERVER-BLINDED STUDY TO EVALUATE THE IMMUNOGENICITY, SAFETY, AND TOLERABILITY OF 2 DOSES COMPARED TO 3 DOSES OF CLOSTRIDIUM DIFFICILE VACCINE IN ADULTS 50 YEARS OF AGE AND OLDER
Brief Title: Clostridium Difficile Vaccine 2-Dose Versus 3-Dose Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B5091019
Record Dates: First submitted 2019-04-02; First posted 2019-04-17 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Clostridium Difficile Associated Disease
Keywords: Clostridium Difficile; vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clostridium difficile vaccine - 3 dose (Experimental): All 3 doses are the Clostridium difficile vaccine
  Interventions: Biological: Clostridium difficile
- Clostridium difficile vaccine - 2 dose (Experimental): 2 of the 3 doses are the Clostridium difficile vaccine with the other being placebo
  Interventions: Biological: Clostridium difficile; Biological: Placebo

INTERVENTIONS:
Biological: Clostridium difficile — Toxoid-based Clostridium difficile vaccine
Biological: Placebo — Normal saline solution (0.9% sodium chloride)
  Arms: Clostridium difficile vaccine - 2 dose

SUMMARY:
This study will investigate a Clostridium difficile vaccine in adults 50 years of age and older. In half the adults, all 3 doses given are the Clostridium difficile vaccine, and in half the adults, 2 of the 3 doses are the Clostridium difficile vaccine with the other dose containing no active ingredients. The study will look at the subjects' immune response to the vaccine and assess the safety and tolerability of a 2-dose regimen of Clostridium difficile vaccine compared to a 3-dose regimen of Clostridium difficile vaccine.

DETAILED DESCRIPTION:
Serology for B5091019 will be forthcoming. There have been delays due to discussions with the FDA on statistical analysis as well as delays attributable to the COVID pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document.
* Willing and able to comply with study procedures.
* Subjects with an increased risk of future contact with healthcare systems or subjects who have received systemic antibiotics in the previous 12 weeks.
* Ability to be contacted by telephone during study participation.

Exclusion Criteria:

* Pregnant female participants; breastfeeding female participants; positive urine pregnancy test for women of childbearing potential (WOCBP); and WOCBP who are, in the opinion of the investigator, sexually active and at risk for pregnancy and are unwilling or unable to use effective methods of contraception as outlined in this protocol from the signing of the informed consent until at least 28 days after the last dose of investigational product.
* Prior episode of CDI, confirmed by either laboratory test or diagnosis of pseudomembranous colitis at colonoscopy, at surgery, or histopathologically.
* Participants who may be unable to respond to vaccination due to:

  * Metastatic malignancy; or
  * End-stage renal disease (glomerular filtration rate <15 mL/min/1.73 m2 or on dialysis).
  * Any serious medical disorder that in the investigator's opinion is likely to be fatal within the next 12 months.
  * Congenital or acquired immunodeficiency.
* Known infection with human immunodeficiency virus (HIV).
* Any bleeding disorder or anticoagulant therapy that would contraindicate IM injection.
* Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Previous administration of an investigational C difficile vaccine or C difficile mAb therapy.
* Receipt of systemic corticosteroids for greater than or equal to 14 days within 28 days before enrollment.
* Receipt of chronic systemic treatment with other known immunosuppressant medications, or radiotherapy, within 6 months before enrollment.
* Receipt of blood products or immunoglobulins within 6 months before enrollment.
* Participation in other studies involving investigational drug(s)/vaccine(s) within 28 days prior to study entry until 1 month after the third vaccination.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1994 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (50):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - East Valley Gastroenterology and Hepatology Associates, Chandler, Arizona
  - The Pain Center of Arizona, Peoria, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Paradigm Clinical Research Centers, Inc., La Mesa, California
  - Paradigm Clinical Research Centers, Inc., Redding, California
  - Paradigm Research, Wheat Ridge, Colorado
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Pines Care Research Center, LLC, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - MOC Research, Mishawaka, Indiana
  - MedPharmics, LLC, Metairie, Louisiana
  - MedPharmics, LLC, Gulfport, Mississippi
  - Clinical Research Professionals Inc., Chesterfield, Missouri
  - Amici Clinical Research, Raritan, New Jersey
  - Rochester Clinical Research, Inc, Rochester, New York
  - PMG Research of Charlotte LLC, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Accellacare - Hickory, Hickory, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Aventiv Research Inc., Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Medical Research South, Goose Creek, South Carolina
  - Main Street Physician's Care - Waterway, Little River, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - ARC Clinical Research at Wilson Parke, Austin, Texas
  - Bellaire Doctor's Clinic, Bellaire, Texas
  - Texas Health Care, PLLC, Fort Worth, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research Inc. / Foothill Family Clinic Draper, Draper, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
  - Virginia Research Center LLC, Midlothian, Virginia
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5091019

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2160 participants signed the inform consent form (ICF).166 participants were screen failures who did not meet criteria and were not enrolled. 1994 participants were randomized, and 1991 participants received study treatment.
Groups:
- 2-Dose Clostridium Difficile Vaccine: Participants received 1 dose of toxin-based Clostridium difficile vaccine intramuscularly at visit 1 (Month 0) and visit 4 (Month 6) and 1 dose of placebo (0.9% sodium chloride) at visit 2 (Month 1). Participants were followed up to 6 months after last dose of vaccination at Month 6.
- 3-Dose Clostridium Difficile Vaccine: Participants were randomized to receive 1 dose of toxin-based Clostridium difficile vaccine intramuscularly at visit 1 (Month 0), visit 2 (Month 1), and visit 4 (Month 6). Participants were followed up to 6 months after last dose of vaccination at Month 6.
Period: Overall Study
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Started | 996 | 998
Vaccinated With Dose 1 | 994 | 997
Vaccinated With Dose 2 | 961 | 964
Vaccinated With Dose 3 | 897 | 917
Completed | 863 | 880
Not Completed | 133 | 118
Not completed — Adverse Event | 19 | 20
Not completed — Death | 14 | 7
Not completed — Lost to Follow-up | 36 | 28
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 7 | 4
Not completed — Withdrawal by Subject | 47 | 47
Not completed — Other | 7 | 11
Not completed — Randomized but not vaccinated | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of the investigational product.
Groups:
- 3-Dose Clostridium Difficile Vaccine: Participants received 1 dose of toxin-based Clostridium difficile vaccine intramuscularly at visit 1 (Month 0), visit 2 (Month 1), and visit 4 (Month 6). Participants were followed up to 6 months after last dose of vaccination at Month 6.
- Total: Total of all reporting groups
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine | Total
Number analyzed (Participants) | 994 | 997 | 1991
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (7.6) | 67.8 (7.5) | 67.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 583 | 598 | 1181
  Male | 411 | 399 | 810
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 113 | 89 | 202
  Not Hispanic or Latino | 869 | 889 | 1758
  Unknown or Not Reported | 12 | 19 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 88 | 90 | 178
  White | 893 | 892 | 1785
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Mean Concentration (GMC) of Clostridium Difficile Toxin A and Toxin B Specific Neutralizing Antibodies at Month 7 for Evaluable Immunogenicity Population (EIP)
Description: Adjusted GMCs and 2-sided 95% confidence intervals (CIs) of toxin A and toxin B specific neutralizing antibody levels were calculated by exponentiating the least square (LS) means and the corresponding CIs based on analysis of logarithmically transformed concentrations using a linear regression model with terms of baseline concentration (log scale) and vaccine group. EIP at Month 7 (EI7): all enrolled participants who received all 3 doses of investigational product; had blood drawn for assay testing within 28 to 47 days after visit 4; had valid and determinate assay results for either toxin A or B for the specified analysis at Month 7; had no major protocol deviations.
Time Frame: Month 7
Population: EI7 population. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" signifies participants with valid and determinate assay results for the specified assay at both baseline and the given sampling time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Neutralization units per milliliter
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 795 | 812
Neutralization units per milliliter
  Toxin A: number analyzed (Participants) | 790 | 805
  Toxin A | 693.0 [646.5 to 742.9] | 845.7 [789.5 to 906.0]
  Toxin B: number analyzed (Participants) | 794 | 810
  Toxin B | 4166.2 [3759.7 to 4616.7] | 7342.9 [6633.1 to 8128.5]
Statistical Analysis 1: Comparison: 2-Dose Clostridium Difficile Vaccine vs 3-Dose Clostridium Difficile Vaccine; Toxin A; Test type: Non-Inferiority — The noninferiority objective was achieved if the lower limit of the 95% CI for geometric mean ratio (GMR) was >0.67 for both Toxin A and Toxin B; Adjusted Geometric Mean Ratio = 0.82, 95% CI 2-sided [0.74 to 0.90] — Adjusted geometric mean ratio (GMR) was estimated by the ratio of the adjusted GMCs (adjusted for baseline concentrations). CIs based on the student t distribution for the mean or the mean difference in logarithmic scale
Statistical Analysis 2: Comparison: 2-Dose Clostridium Difficile Vaccine vs 3-Dose Clostridium Difficile Vaccine; Toxin B; Test type: Non-Inferiority — The noninferiority objective was achieved if the lower limit of the 95% CI for GMR was >0.67 for both Toxin A and Toxin B; Adjusted Geometric Mean Ratio = 0.57, 95% CI 2-sided [0.49 to 0.66] — Adjusted GMR was estimated by the ratio of the adjusted GMCs (adjusted for baseline concentrations). CIs based on the student t distribution for the mean difference in logarithmic scale

2. Primary Outcome: Percentage of Participants Achieving Seroresponse for Clostridium Difficile Toxin A and Toxin B at Month 7 for EIP
Description: Seroresponse was defined as at least a 4-fold rise from the baseline neutralizing antibody level following vaccination. 95% CI was based on Clopper-Pearson method. EI7: all enrolled participants who received all 3 doses of investigational product; had blood drawn for assay testing within 28 to 47 days after visit 4; had valid and determinate assay results for either toxin A or B for the specified analysis at Month 7; had no major protocol deviations.
Time Frame: Month 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 795 | 812
Percentage of participants
  Toxin A: number analyzed (Participants) | 790 | 805
  Toxin A | 32.2 [28.9 to 35.5] | 33.9 [30.6 to 37.3]
  Toxin B: number analyzed (Participants) | 794 | 810
  Toxin B | 56.7 [53.1 to 60.2] | 73.5 [70.3 to 76.5]
Statistical Analysis 1: Comparison: 2-Dose Clostridium Difficile Vaccine vs 3-Dose Clostridium Difficile Vaccine; Toxin A; Test type: Non-Inferiority — The noninferiority objective was achieved if the lower limit of the 95% CI for the difference was >-10% for both Toxin A and Toxin B; Percentage difference = -1.8, 95% CI 2-sided [-6.4 to 2.9] — The difference (2-Dose - 3-Dose) and the associated 95% CIs for the difference were calculated using the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: 2-Dose Clostridium Difficile Vaccine vs 3-Dose Clostridium Difficile Vaccine; Toxin B; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage difference = -16.8, 95% CI 2-sided [-21.3 to -12.2] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Percentage of Participants With Local Reactions by Maximum Severity Through 7 Days After Dose 1
Description: Local reactions included pain at injection site, redness and swelling. These were recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit= 0.5 centimeter (cm). Redness and swelling were graded as mild: 2.5-5.0 cm, moderate: greater than (>) 5.0-10.0 cm, severe: >10.0 cm, potentially life threatening: necrosis or exfoliative dermatitis for redness, or necrosis for swelling. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity, potentially life threatening: emergency room visit or hospitalization. The maximum severity was defined as highest grading of each local reaction through 7 days of vaccination.
Time Frame: Up to 7 days after Dose 1 of investigational product at Month 0
Population: Safety analysis set included all participants who received at least 1 dose of the investigational product. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 983 | 988
Percentage of participants
  Pain at injection site: Mild | 19.1 [16.7 to 21.7] | 17.5 [15.2 to 20.0]
  Pain at injection site: Moderate | 1.2 [0.6 to 2.1] | 2.6 [1.7 to 3.8]
  Pain at injection site: Severe | 0.0 [0.0 to 0.4] | 0.1 [0.0 to 0.6]
  Pain at injection site: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Redness: Mild | 0.9 [0.4 to 1.7] | 0.6 [0.2 to 1.3]
  Redness: Moderate | 0.2 [0.0 to 0.7] | 0.6 [0.2 to 1.3]
  Redness: Severe | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Redness: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Swelling: Mild | 1.9 [1.2 to 3.0] | 1.6 [0.9 to 2.6]
  Swelling: Moderate | 0.7 [0.3 to 1.5] | 0.8 [0.4 to 1.6]
  Swelling: Severe | 0.0 [0.0 to 0.4] | 0.1 [0.0 to 0.6]
  Swelling: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]

4. Primary Outcome: Percentage of Participants With Local Reactions by Maximum Severity Through 7 Days After Dose 2
Description: Local reactions included pain at injection site, redness and swelling. These were recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit= 0.5 cm. Redness and swelling were graded as mild: 2.5-5.0 cm, moderate: >5.0-10.0 cm, severe: >10.0 cm, potentially life threatening: necrosis or exfoliative dermatitis for redness, or necrosis for swelling. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity, potentially life threatening: emergency room visit or hospitalization. The maximum severity was defined as highest grading of each local reaction through 7 days of vaccination.
Time Frame: Up to 7 days after Dose 2 of investigational product at Month 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 937 | 940
Percentage of participants
  Pain at injection site: Mild | 5.4 [4.1 to 7.1] | 24.0 [21.3 to 26.9]
  Pain at injection site: Moderate | 0.4 [0.1 to 1.1] | 4.0 [2.9 to 5.5]
  Pain at injection site: Severe | 0.2 [0.0 to 0.8] | 0.4 [0.1 to 1.1]
  Pain at injection site: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Redness: Mild | 0.0 [0.0 to 0.4] | 2.3 [1.5 to 3.5]
  Redness: Moderate | 0.2 [0.0 to 0.8] | 1.6 [0.9 to 2.6]
  Redness: Severe | 0.0 [0.0 to 0.4] | 0.5 [0.2 to 1.2]
  Redness: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Swelling: Mild | 0.6 [0.2 to 1.4] | 3.5 [2.4 to 4.9]
  Swelling: Moderate | 0.3 [0.1 to 0.9] | 3.2 [2.2 to 4.5]
  Swelling: Severe | 0.1 [0.0 to 0.6] | 0.5 [0.2 to 1.2]
  Swelling: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]

5. Primary Outcome: Percentage of Participants With Local Reactions by Maximum Severity Through 7 Days After Dose 3
Description: as for outcome 4
Time Frame: Up to 7 days after Dose 3 of investigational product at Month 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 869 | 894
Percentage of participants
  Pain at injection site: Mild | 23.7 [20.9 to 26.7] | 23.5 [20.7 to 26.4]
  Pain at injection site: Moderate | 5.2 [3.8 to 6.9] | 4.9 [3.6 to 6.6]
  Pain at injection site: Severe | 0.2 [0.0 to 0.8] | 0.1 [0.0 to 0.6]
  Pain at injection site: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Redness: Mild | 2.5 [1.6 to 3.8] | 2.8 [1.8 to 4.1]
  Redness: Moderate | 2.2 [1.3 to 3.4] | 2.1 [1.3 to 3.3]
  Redness: Severe | 0.0 [0.0 to 0.4] | 0.3 [0.1 to 1.0]
  Redness: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Swelling: Mild | 3.3 [2.2 to 4.8] | 4.8 [3.5 to 6.4]
  Swelling: Moderate | 3.3 [2.2 to 4.8] | 2.6 [1.6 to 3.8]
  Swelling: Severe | 0.2 [0.0 to 0.8] | 0.3 [0.1 to 1.0]
  Swelling: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]

6. Primary Outcome: Percentage of Participants With Systemic Events by Maximum Severity Through 7 Days After Dose 1
Description: Systemic events included fever, fatigue, headache, joint pain, muscle pain and vomiting. These were recorded by participants in an e-diary. Fever was categorized as: mild (38.0 to 38.4 degree [deg] Celsius [C]), moderate (38.5 to 38.9 deg C), severe (39.0 to 40.0 deg C) and potentially life threatening (>40.0 deg C). Fatigue, headache, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity, severe: prevented daily routine activity and potentially life threatening: emergency room visit or hospitalization. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h, severe: required intravenous hydration and potentially life threatening: emergency room visit or hospitalization for hypotensive shock. The maximum severity was defined as highest grading of each systemic event through 7 days of vaccination.
Time Frame: Up to 7 days after Dose 1 of investigational product at Month 0
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 983 | 988
Percentage of participants
  Fever: 38.0-38.4 deg C | 0.5 [0.2 to 1.2] | 0.9 [0.4 to 1.7]
  Fever: 38.5-38.9 deg C | 0.2 [0.0 to 0.7] | 0.1 [0.0 to 0.6]
  Fever: 39.0-40.0 deg C | 0.0 [0.0 to 0.4] | 0.1 [0.0 to 0.6]
  Fever: >40.0 deg C | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Fatigue: Mild | 11.3 [9.4 to 13.4] | 14.1 [12.0 to 16.4]
  Fatigue: Moderate | 14.6 [12.5 to 17.0] | 15.5 [13.3 to 17.9]
  Fatigue: Severe | 1.9 [1.2 to 3.0] | 1.8 [1.1 to 2.9]
  Fatigue: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Headache: Mild | 13.5 [11.5 to 15.8] | 14.5 [12.3 to 16.8]
  Headache: Moderate | 7.5 [6.0 to 9.4] | 8.2 [6.6 to 10.1]
  Headache: Severe | 0.4 [0.1 to 1.0] | 0.4 [0.1 to 1.0]
  Headache: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Joint pain: Mild | 4.9 [3.6 to 6.4] | 5.2 [3.9 to 6.7]
  Joint pain: Moderate | 5.6 [4.2 to 7.2] | 5.2 [3.9 to 6.7]
  Joint pain: Severe | 0.6 [0.2 to 1.3] | 0.1 [0.0 to 0.6]
  Joint pain: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Muscle pain: Mild | 5.6 [4.2 to 7.2] | 5.1 [3.8 to 6.6]
  Muscle pain: Moderate | 6.5 [5.0 to 8.2] | 7.4 [5.8 to 9.2]
  Muscle pain: Severe | 1.0 [0.5 to 1.9] | 0.5 [0.2 to 1.2]
  Muscle pain: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Vomiting: Mild | 1.2 [0.6 to 2.1] | 1.9 [1.2 to 3.0]
  Vomiting: Moderate | 0.2 [0.0 to 0.7] | 0.4 [0.1 to 1.0]
  Vomiting: Severe | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Vomiting: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]

7. Primary Outcome: Percentage of Participants With Systemic Events by Maximum Severity Through 7 Days After Dose 2
Description: Systemic events included fever, fatigue, headache, joint pain, muscle pain and vomiting. These were recorded by participants in an e-diary. Fever was categorized as: mild (38.0 to 38.4 deg C), moderate (38.5 to 38.9 deg C), severe (39.0 to 40.0 deg C) and potentially life threatening (>40.0 deg C). Fatigue, headache, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity, severe: prevented daily routine activity and potentially life threatening: emergency room visit or hospitalization. Vomiting was graded as mild: 1 to 2 times in 24h, moderate: >2 times in 24h, severe: required intravenous hydration and potentially life threatening: emergency room visit or hospitalization for hypotensive shock. The maximum severity was defined as highest grading of each systemic event through 7 days of vaccination.
Time Frame: Up to 7 days after Dose 2 of investigational product at Month 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 937 | 940
Percentage of participants
  Fever: 38.0-38.4 deg C | 0.6 [0.2 to 1.4] | 0.3 [0.1 to 0.9]
  Fever: 38.5-38.9 deg C | 0.3 [0.1 to 0.9] | 0.3 [0.1 to 0.9]
  Fever: 39.0-40.0 deg C | 0.1 [0.0 to 0.6] | 0.2 [0.0 to 0.8]
  Fever: >40.0 deg C | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Fatigue: Mild | 9.5 [7.7 to 11.6] | 12.1 [10.1 to 14.4]
  Fatigue: Moderate | 11.2 [9.3 to 13.4] | 12.6 [10.5 to 14.8]
  Fatigue: Severe | 1.3 [0.7 to 2.2] | 1.6 [0.9 to 2.6]
  Fatigue: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Headache: Mild | 9.8 [8.0 to 11.9] | 10.9 [8.9 to 13.0]
  Headache: Moderate | 6.1 [4.6 to 7.8] | 7.8 [6.1 to 9.7]
  Headache: Severe | 0.7 [0.3 to 1.5] | 0.7 [0.3 to 1.5]
  Headache: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Joint pain: Mild | 2.0 [1.2 to 3.1] | 2.6 [1.6 to 3.8]
  Joint pain: Moderate | 4.8 [3.5 to 6.4] | 5.6 [4.3 to 7.3]
  Joint pain: Severe | 0.6 [0.2 to 1.4] | 1.0 [0.4 to 1.8]
  Joint pain: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Muscle pain: Mild | 3.2 [2.2 to 4.5] | 3.6 [2.5 to 5.0]
  Muscle pain: Moderate | 5.2 [3.9 to 6.9] | 7.7 [6.0 to 9.5]
  Muscle pain: Severe | 0.6 [0.2 to 1.4] | 0.7 [0.3 to 1.5]
  Muscle pain: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Vomiting: Mild | 0.9 [0.4 to 1.7] | 0.9 [0.4 to 1.7]
  Vomiting: Moderate | 0.5 [0.2 to 1.2] | 0.4 [0.1 to 1.1]
  Vomiting: Severe | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Vomiting: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]

8. Primary Outcome: Percentage of Participants With Systemic Events by Maximum Severity Through 7 Days After Dose 3
Description: as for outcome 7
Time Frame: Up to 7 days after Dose 3 of investigational product at Month 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 869 | 894
Percentage of participants
  Fever: 38.0-38.4 deg C | 0.3 [0.1 to 1.0] | 0.1 [0.0 to 0.6]
  Fever: 38.5-38.9 deg C | 0.0 [0.0 to 0.4] | 0.1 [0.0 to 0.6]
  Fever: 39.0-40.0 deg C | 0.3 [0.1 to 1.0] | 0.0 [0.0 to 0.4]
  Fever: >40.0 deg C | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Fatigue: Mild | 9.1 [7.3 to 11.2] | 9.6 [7.8 to 11.7]
  Fatigue: Moderate | 11.3 [9.3 to 13.6] | 13.1 [10.9 to 15.5]
  Fatigue: Severe | 1.6 [0.9 to 2.7] | 0.9 [0.4 to 1.8]
  Fatigue: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Headache: Mild | 11.5 [9.5 to 13.8] | 12.8 [10.6 to 15.1]
  Headache: Moderate | 7.6 [5.9 to 9.6] | 5.1 [3.8 to 6.8]
  Headache: Severe | 0.7 [0.3 to 1.5] | 0.7 [0.2 to 1.5]
  Headache: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Joint pain: Mild | 2.9 [1.9 to 4.2] | 2.6 [1.6 to 3.8]
  Joint pain: Moderate | 5.2 [3.8 to 6.9] | 3.6 [2.5 to 5.0]
  Joint pain: Severe | 0.3 [0.1 to 1.0] | 0.2 [0.0 to 0.8]
  Joint pain: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Muscle pain: Mild | 5.5 [4.1 to 7.3] | 4.8 [3.5 to 6.4]
  Muscle pain: Moderate | 6.2 [4.7 to 8.0] | 4.9 [3.6 to 6.6]
  Muscle pain: Severe | 0.1 [0.0 to 0.6] | 0.3 [0.1 to 1.0]
  Muscle pain: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Vomiting: Mild | 1.2 [0.6 to 2.1] | 1.5 [0.8 to 2.5]
  Vomiting: Moderate | 0.5 [0.1 to 1.2] | 0.2 [0.0 to 0.8]
  Vomiting: Severe | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Vomiting: Potentially life threatening | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]

9. Primary Outcome: Percentage of Participants With Adverse Events Through 1 Month After Last Study Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Percentage of participants with any AEs (both serious and all non-serious AEs) and non-serious AEs through 1 month after last study vaccination were reported in this outcome measure. Only AEs and non-SAEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From day of first dose up to 1 month after last dose (up to Month 7)
Population: Safety analysis set included all participants who received at least 1 dose of the investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 994 | 997
Percentage of participants
  Any AEs | 47.7 | 49.7
  Non-Serious AEs | 44.8 | 46.8

10. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Through 6 Months After Last Study Vaccination
Description: SAE was any untoward medical occurrence that at any dose resulted in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From day of first dose up to 6 months after last dose (up to Month 12)
Population: Safety analysis set included all participants who received at least 1 dose of the investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 994 | 997
Percentage of participants | 14.2 | 13.6

11. Secondary Outcome: Adjusted Geometric Mean Concentration for Clostridium Difficile Toxin A and Toxin B Specific Neutralizing Antibody at Month 12 for EIP
Description: Adjusted GMCs and 2-sided 95% CIs of toxin A and toxin B specific neutralizing antibody levels were calculated by exponentiating the LS means and the corresponding CIs based on analysis of logarithmically transformed concentrations using a linear regression model with terms of baseline concentration (log scale) and vaccine group. EI12: all enrolled participants who received all 3 doses of investigational product; had blood drawn for assay testing within 165 to 200 days after visit 4; had valid and determinate assay results for either toxin A or B for the specified analysis at Month 12; had no major protocol deviations.
Time Frame: Month 12
Population: EI12 population. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" signifies participants with valid and determinate assay results for the specified assay at both baseline and the given sampling time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Neutralization units per milliliter
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 801 | 825
Neutralization units per milliliter
  Toxin A: number analyzed (Participants) | 800 | 822
  Toxin A | 327.5 [307.9 to 348.3] | 375.5 [353.4 to 399.1]
  Toxin B: number analyzed (Participants) | 801 | 824
  Toxin B | 2230.8 [2033.9 to 2446.7] | 3149.8 [2875.5 to 3450.1]
Statistical Analysis 1: Comparison: 2-Dose Clostridium Difficile Vaccine vs 3-Dose Clostridium Difficile Vaccine; Toxin A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Adjusted Geometric Mean Ratio = 0.87, 95% CI 2-sided [0.80 to 0.95] — Adjusted GMR was estimated by the ratio of the adjusted GMCs (adjusted for baseline concentrations). CIs based on the student t distribution for the mean or the mean difference in logarithmic scale
Statistical Analysis 2: Comparison: 2-Dose Clostridium Difficile Vaccine vs 3-Dose Clostridium Difficile Vaccine; Toxin B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Adjusted Geometric Mean Ratio = 0.71, 95% CI 2-sided [0.62 to 0.81] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Percentage of Participants Achieving Seroresponse for Clostridium Difficile Toxin A and Toxin B at Month 12 for EIP
Description: Seroresponse was defined as at least a 4-fold rise from the baseline neutralizing antibody following vaccination. 95% CI was based on Clopper-Pearson method. EI12: all enrolled participants who received all 3 doses of investigational product; had blood drawn for assay testing within 165 to 200 days after visit 4; had valid and determinate assay results for either toxin A or B for the specified analysis at Month 12; had no major protocol deviations.
Time Frame: Month 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
Number analyzed (Participants) | 801 | 825
Percentage of participants
  Toxin A: number analyzed (Participants) | 800 | 822
  Toxin A | 7.8 [6.0 to 9.8] | 8.8 [6.9 to 10.9]
  Toxin B: number analyzed (Participants) | 801 | 824
  Toxin B | 40.0 [36.5 to 43.4] | 50.2 [46.8 to 53.7]
Statistical Analysis 1: Comparison: 2-Dose Clostridium Difficile Vaccine vs 3-Dose Clostridium Difficile Vaccine; Toxin A; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage difference = -1.0, 95% CI 2-sided [-3.7 to 1.7] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 2-Dose Clostridium Difficile Vaccine vs 3-Dose Clostridium Difficile Vaccine; Toxin B; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage difference = -10.3, 95% CI 2-sided [-15.1 to -5.5] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events: within 7 days after vaccination (systematic assessment), other AEs: from Day 1 up to 1 month after last dose of vaccination (up to Month 7), all-cause mortality and SAEs: from Day 1 up to 6 months after last dose of vaccination (up to Month 12)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety set was evaluated.
Arm/Group | 2-Dose Clostridium Difficile Vaccine | 3-Dose Clostridium Difficile Vaccine
All-Cause Mortality (participants affected / at risk) | 15/994 | 7/997
Serious Adverse Events (participants affected / at risk) | 141/994 | 136/997
Other Adverse Events (participants affected / at risk) | 721/994 | 751/997
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2-Dose Clostridium Difficile Vaccine (N=994) | 3-Dose Clostridium Difficile Vaccine (N=997)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 4
Angina unstable (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 7 | 3
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 6 | 8
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 5 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Familial amyloidosis (Congenital, familial and genetic disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal vascular ectasia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 2 | 8
Death (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 3
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 9
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 2
Epididymitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Metapneumovirus pneumonia (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 10
Pneumonia aspiration (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 7
Septic shock (Infections and infestations) | 0 | 3
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 4
Urosepsis (Infections and infestations) | 1 | 2
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bell's palsy (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Encephalopathy (Nervous system disorders) | 0 | 3
Essential tremor (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 2 | 1
Intracranial mass (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 2
Lacunar infarction (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 3
Nerve compression (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 6 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 1
Tremor (Nervous system disorders) | 0 | 1
Device dislocation (Product Issues) | 0 | 1
Device occlusion (Product Issues) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Behaviour disorder (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Drug abuse (Psychiatric disorders) | 0 | 1
Homicidal ideation (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 7
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1
Hypertensive nephropathy (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal injury (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 1
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Multiple drug therapy (Surgical and medical procedures) | 1 | 0
Oesophagogastric fundoplasty (Surgical and medical procedures) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 2 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2-Dose Clostridium Difficile Vaccine (N=994) | 3-Dose Clostridium Difficile Vaccine (N=997)
Diarrhoea (Gastrointestinal disorders) | 18 | 21
Nausea (Gastrointestinal disorders) | 12 | 14
Vomiting (VOMITING) (Gastrointestinal disorders) | 37 | 45
Fatigue (General disorders) | 13 | 5
Fatigue (FATIGUE) (General disorders) | 426 | 461
Injection site erythema (REDNESS) (General disorders) | 53 | 85
Injection site pain (PAIN) (General disorders) | 378 | 440
Injection site swelling (SWELLING) (General disorders) | 80 | 129
Pyrexia (FEVER) (General disorders) | 23 | 19
Bronchitis (Infections and infestations) | 19 | 9
Cellulitis (Infections and infestations) | 12 | 12
Nasopharyngitis (Infections and infestations) | 15 | 18
Sinusitis (Infections and infestations) | 20 | 25
Upper respiratory tract infection (Infections and infestations) | 44 | 40
Urinary tract infection (Infections and infestations) | 38 | 41
Fall (Injury, poisoning and procedural complications) | 38 | 38
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 24
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 192 | 183
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 14
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 233 | 245
Headache (Nervous system disorders) | 8 | 18
Headache (HEADACHE) (Nervous system disorders) | 359 | 388
Hypertension (Vascular disorders) | 11 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT03918629/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT03918629/SAP_001.pdf